CLINICAL TRIAL: NCT03527277
Title: The Effects of Orange Juice Compared With Sugar-sweetened Beverage on Risk Factors and Metabolic Processes Associated With the Development of Cardiovascular Disease and Type 2 Diabetes
Brief Title: Orange Juice And Sugar Intervention Study
Acronym: OASIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Touro University, California (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kimber Stanhope, Research Nutritional Biologist, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1167030; R01HL137716 (NIH)
Record Dates: First submitted 2018-04-10; First posted 2018-05-17 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Risk Factor; Type2 Diabetes Mellitus; Insulin Sensitivity; Metabolic Syndrome
Keywords: orange juice; sugar-sweetened beverage; triglyceride; low density lipoprotein cholesterol; apolipoprotein B; uric acid; de novo lipogenesis; hepatic triglyceride; hepatic glucose production; whole body insulin sensitivity
MeSH Terms: conditions — Insulin Resistance; Metabolic Syndrome | interventions — Sugar-Sweetened Beverages

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: All outcomes will be analyzed/assessed by subject identity number, which are assigned prior to randomization to experimental arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naturally-sweetened orange juice (Experimental): Naturally-sweetened orange juice Form: Beverage Daily dosage: 25% of daily energy requirement Frequency: Divided into 3 servings/day Duration: 4 weeks
  Interventions: Other: Naturally-sweetened orange juice
- Sugar-sweetened beverage (Active Comparator): Sugar-sweetened beverage Form: Beverage Daily dosage: 25% of daily energy requirement Frequency: Divided into 3 servings/day Duration: 4 weeks
  Interventions: Other: Sugar-sweetened beverage

INTERVENTIONS:
Other: Naturally-sweetened orange juice — Commercially-available ready-to-serve refrigerated orange juice
  Arms: Naturally-sweetened orange juice
Other: Sugar-sweetened beverage — Sugar-sweetened water flavored with Kool-Aid (TM)
  Arms: Sugar-sweetened beverage

SUMMARY:
The objectives of this proposal are to address the gaps in knowledge regarding the metabolic effects of consuming orange juice, the most frequently consumed fruit juice in this country, compared to sugar-sweetened beverage.

DETAILED DESCRIPTION:
Specific Aims: There is considerable epidemiological evidence that demonstrates associations between added sugar/sugar-sweetened beverage consumption and increased risk for or prevalence of chronic diseases such as cardiovascular disease (CVD), type 2 diabetes (T2D), metabolic syndrome, and gout. Especially concerning is recent evidence from National Health and Nutrition Examination Survey III that demonstrates that there is increased risk of CVD mortality with increased intake of added sugar across quintiles (Yang, 2014). Even the US mean added sugar intake, 15% of daily calories, was associated with an 18% increase in risk of CVD mortality over 15 years. The results from the investigator's recently completed study (1R01 HL09133) corroborate these findings (Stanhope, 2015). They demonstrate that supplementing the ad libitum diets of young adults with beverages containing 0, 10, 17.5 or 25% of daily energy requirement (Ereq) as high fructose corn syrup (HFCS) affects lipid/lipoprotein risk factors for CVD in a dose response manner. Specifically, levels of nonHDL-cholesterol(C), LDL-C, apolipoprotein B (apoB), and postprandial triglycerides (TG) increased linearly over a 2-week period with increasing doses of HFCS. Furthermore, even the participants consuming the 10% Ereq dose exhibited increased levels of these risk factors compared to baseline.

These and similar results have helped to lead to reductions in soda consumption in this country, and new dietary guidelines and FDA food labeling requirements to promote reductions in added sugar consumption. However, there are gaps in knowledge about other sugar-containing foods that lead to public confusion concerning healthier options for soda, and impede further progress in implementing public health policies that will promote further reductions in soda consumption. One such food is naturally-sweetened fruit juice. The amount of sugar in fruit juice is comparable to the amount in soda. Because of this, a consumer seeking answers on the internet will find many articles in which experts state or suggest that the effects of consuming fruit juice are as detrimental as or even worse than those of soda. However, in contrast to soda, fruit juice contains micronutrients and bioactives that may promote health. Therefore the consumer can also find numerous articles on the internet where the health benefits of fruit juice and these bioactives are extolled. There are a limited number of clinical dietary intervention studies that have directly compared the metabolic effects of consuming fruit juice and sugar-sweetened beverage, and their results are not conclusive. Thus we will pursue the following Specific Aims:

1. Specific Aim 1: To compare the weight-independent effects of consuming 25%Ereq as orange juice or sugar-sweetened beverages for 4 weeks on risk factors for CVD and other chronic disease in normal weight and overweight men and women.
2. Specific Aim 2: To mechanistically compare the weight-independent effects of consuming 25%Ereq as orange juice or sugar-sweetened beverages on metabolic processes associated with the development of CVD and T2D in normal weight and overweight men and women.
3. Specific Aim 3: To relate the changes assessed under Specific Aims 1 and 2 to the changes in the urinary levels of metabolites and catabolites of the main flavanones in orange juice, hesperetin and naringenin.

ELIGIBILITY:
Inclusion Criteria: men and pre-menopausal women Body mass index: 20-35 kg/m2 Body weight > than 50 kg Self-reported stable body weight during the prior six months

Exclusion Criteria:

Fasting glucose >125 mg/dl Evidence of liver disorder (AST or ALT >200% upper limit of normal range) Evidence of kidney disorder (>2.0 mg/dl creatinine) Evidence of thyroid disorder (out of normal range) Systolic blood pressure consistently over 140 mmHg or diastolic blood pressure over 90 mmHg Triglycerides > 400 mg/dl LDL-C > 160 mg/dl in combination with Chol:HDL > 4 Hemoglobin < 10 g/dL Pregnant or lactating women Current, prior (within 12 months), or anticipated use of any hypolipidemic or anti-diabetic agents.

Use of thyroid, anti-hypertensive, anti-depressant, weight loss medications or any other medication which, in the opinion of the investigator, may confound study results Use of tobacco Strenuous exerciser (>3.5 hours/week at a level more vigorous than walking) Surgery for weight loss Diet exclusions: Food allergies, special dietary restrictions, routine consumption of less than 3 meals/day, routine ingestion of more than 2 sugar-sweetened beverages or 1 alcoholic beverage/day, unwillingness to consume any food on study menu Veins that are assessed by the R.N.s as being unsuitable for long-term infusions and multiple blood draws from a catheter.

Pre-existing claustrophobia or metal implants that preclude magnetic resonance imaging Any other condition that, in the opinion of the investigators, would put the subject at risk

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self-representation
Enrollment: 56 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2023-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimber L Stanhope, Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Final dataset will include data collected specifically for the study and data provided during screening in the medical history form. This includes some demographic information and data regarding family history of disease. We will make data and demographic information available to other investigators upon request. The dataset will be stripped of all unique identifiers and subject characteristics and prepared in accordance with all HIPAA regulations prior to release for sharing. Study outcome results will be submitted to ClinicalTrials.gov no later than one year after the trial's primary completion date.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after the end of study--January 31, 2025
Access Criteria: We will make data and demographic information available to investigators who submit an outline with:
  1. Hypotheses/aims
  2. Assurance that the data will be stored on secured computer
  3. Assurance that access will be limited to those named in the proposal
  4. Commitment to destroy/return the data after analyses are completed
  5. Guarantee that the grant and the primary investigators will be acknowledged in any publications arising from these data.

REFERENCES:
- [Result] Yang Q, Zhang Z, Gregg EW, Flanders WD, Merritt R, Hu FB. Added sugar intake and cardiovascular diseases mortality among US adults. JAMA Intern Med. 2014 Apr;174(4):516-24. doi: 10.1001/jamainternmed.2013.13563. PMID 24493081
- [Result] Stanhope KL, Medici V, Bremer AA, Lee V, Lam HD, Nunez MV, Chen GX, Keim NL, Havel PJ. A dose-response study of consuming high-fructose corn syrup-sweetened beverages on lipid/lipoprotein risk factors for cardiovascular disease in young adults. Am J Clin Nutr. 2015 Jun;101(6):1144-54. doi: 10.3945/ajcn.114.100461. Epub 2015 Apr 22. PMID 25904601
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-the-effect-of-orange-juice-or-sugar-sweetened-beverages-on-risk-factors-for-type-2-diabetes-and-cardiovascular-disease-564592/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Started | 31 | 25
Completed | 25 | 24
Not Completed | 6 | 1
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Withdrawn by PI due to veins not suitable for multiple blood draws | 0 | 1
Not completed — Withdrawn by PI due to dietary miscompliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (3.8) | 24.8 (7.1) | 23.8 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 15 | 13 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 16 | 15 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49
Body Mass Index [Mean (Standard Deviation); unit: kg/meters^2] — Body Weight (kg)/(Height (meters))*(Height (meters))
  kg/meters^2 | 23.8 (3.6) | 24.0 (3.3) | 23.9 (3.4)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Systolic blood pressure during fasting (mmHg)
  mmHg | 110.8 (11.0) | 111.0 (11.4) | 110.9 (11.1)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Systolic blood pressure during fasting (mmHg)
  mmHg | 71.0 (7.5) | 69.7 (8.3) | 70.4 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Fasting Low Density Lipoprotein Cholesterol (LDL-C)
Description: Absolute change of plasma LDL-C concentration (4 week value - 0 week value)
Time Frame: 4 weeks
Population: One participant was excluded due to extreme values that deviated from the mean by more than 2 standard deviations across multiple outcomes. The exclusion was based on protocol-defined criteria.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
mg/dl | 5.5 (5.3) | 5.8 (7.5)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.88, ANCOVA; Effect of group on change of outcome with adjustment for BMI, Outcome at baseline and gender; Mean Difference (Net) = -0.3, 95% CI 2-sided [-4.0 to 3.5]

2. Primary Outcome: Postprandial Low Density Lipoprotein Cholesterol (LDL-C)
Description: Absolute change of plasma postprandial LDL-C concentration (4 week value - 0 week value)
Time Frame: 4 weeks
Population: One participant was excluded due to extreme values that deviated from the mean by more than 2 standard deviations across multiple outcomes. The exclusion was based on protocol-defined criteria. Unable to collect week 4 postprandial samples from one participant in the Sucrose Group
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 22
mg/dl | 5.9 (4.8) | 6.7 (5.6)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.65, ANCOVA; Effect of group on change of outcome with adjustment for gender and outcome and BMI at baseline; Mean Difference (Net) = -0.7, 95% CI 2-sided [-3.7 to 2.3]

3. Primary Outcome: Fasting Apolipoprotein B (apoB)
Description: Absolute change of plasma apoB concentration (4 week value - 0 week value)
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
mg/dl | 2.9 (4.6) | 3.4 (7.5)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.92, ANCOVA; Effect of group on change of outcome with adjustment for gender and outcome and BMI at baseline; Mean Difference (Net) = -0.2, 95% CI 2-sided [-3.7 to 3.4]

4. Primary Outcome: Postprandial Apolipoprotein B (apoB)
Description: Absolute change of plasma postprandial apoB concentration (4 week value - 0 week value)
Time Frame: 4 weeks
Population: One participant was excluded due to extreme values that deviated from the mean by more than 2 standard deviations across multiple outcomes. The exclusion was based on protocol-defined criteria. Unable to collect post-dinner blood samples from one participant in the sucrose group during the 4-week intervention trial.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 22
mg/dl | 3.7 (4.5) | 4.3 (5.9)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.81, ANCOVA; Effect of group on change of outcome with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = -0.4, 95% CI 2-sided [-3.3 to 2.6]

5. Primary Outcome: Fasting Uric Acid
Description: Absolute change of plasma uric acid concentration (4 week value - 0 week value)
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
mg/dl | -0.92 (0.85) | 0.11 (0.60)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p < 0.0001, ANCOVA; Effect of group with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = -0.92, 95% CI 2-sided [-1.34 to -0.49]

6. Primary Outcome: Postprandial Uric Acid
Description: Absolute change of post-dinner 4-hour AUC plasma uric acid concentration (4 week value - 0 week value)
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dl x 4 h
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 22
mg/dl x 4 h | -3.3 (2.6) | 0.40 (1.9)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p < 0.0001, ANCOVA; Effect of group on change of outcome with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = -3.4, 95% CI 2-sided [-4.7 to -2.1]

7. Primary Outcome: Fasting Apolipoprotein CIII (apoCIII)
Description: Absolute change of fasting plasma apoCIII concentration (4 week value - 0 week value)
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
mg/dl | 0.40 (1.03) | 0.60 (0.92)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.42, ANCOVA; Effect of group on change of outcome with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.74 to 0.31]

8. Primary Outcome: Postprandial Apolipoprotein CIII (apoCIII)
Description: Absolute change of plasma postprandial apoCIII concentration (4 week value - 0 week value)
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 22
mg/dl | 0.64 (0.93) | 0.38 (0.85)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.28, ANCOVA; Effect of group on change of outcome with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = 0.27, 95% CI 2-sided [-0.23 to 0.76]

9. Primary Outcome: Postprandial Triglyceride
Description: Absolute change of 4-h post-dinner AUC plasma triglyceride concentration (4 week value - 0 week value)
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dl x 4 h
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 22
mg/dl x 4 h | 41.8 (61.3) | 53.5 (56.9)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.59, ANCOVA; Effect of group on change of outcome with adjustment of gender and BMI and outcome at baseline; Mean Difference (Net) = -9.1, 95% CI 2-sided [-42.9 to 24.7]

10. Primary Outcome: Hepatic Triglyceride
Description: Absolute change of % hepatic triglyceride (4 week value - 0 week value)
Time Frame: 4 weeks
Population: One participant was excluded due to extreme values that deviated from the mean by more than 2 standard deviations across multiple outcomes. The exclusion was based on protocol-defined criteria. One participant in the Orange Juice Group was not able to attend the intervention MRI appointment.
Measure: Mean (Standard Deviation); unit: % fat in liver
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 24 | 23
% fat in liver | 0.05 (0.86) | 0.26 (0.53)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.35, ANCOVA; Effect of group on change of outcome with adjustment for gender and outcome at baseline; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.21 to 0.08]

11. Primary Outcome: Matsuda Insulin Sensitivity Index (ISI)
Description: Absolute change of Matsuda ISI (4 week value - 0 week value). The Matsuda Index is a ratio of glucose and insulin levels during oral glucose tolerance test. It is calculated using fasting and mean glucose and insulin measurements, but the units of these measurements cancel out in the formula. A Matsuda value less than 2.5 may indicate insulin resistance, thus a lowering of the Matsuda index is a detrimental outcome.
  At baseline the Matsuda index in the participants for which it was assessed ranged from 1.4 to 7.8 (mean = 3.7, standard deviation = 1.6).
Time Frame: 4 week
Population: This analysis includes participants enrolled after a coronavirus disease 2019 (COVID)-related protocol modification, who completed a 3-hour OGTT. These participants (n=39) did not undergo hyperinsulinemic euglycemic clamps. Final data collection and analysis for this population are complete. One participant was excluded due to extreme values that deviated from the mean by more than 2 standard deviations across multiple outcomes. The exclusion was based on protocol-defined criteria.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 21 | 17
units on a scale | -0.35 (1.0) | -0.40 (0.98)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.97, ANCOVA; Effect of group on change of outcome with adjustment for gender and outcome and BMI at baseline; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.61 to 0.59]

12. Primary Outcome: Postprandial de Novo Lipogenesis
Description: Absolute change of 8-hour area under the curve (AUC) percentage fractional rate postprandial de novo lipogenesis DNL (4 week value - 0 week value)
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: %fractional rate x 8 h
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 22
%fractional rate x 8 h | 8.3 (12.3) | 22.3 (16.2)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Effect of group on change of outcome with adjustment for BMI, outcome at baseline and gender; Test type: Superiority; p = 0.002, ANCOVA; Effect of group on change of outcome with adjustment for gender and outcome and BMI at baseline; Mean Difference (Net) = -13.9, 95% CI 2-sided [-22.4 to -5.4]

13. Secondary Outcome: Fasting Triglyceride
Description: Absolute change of plasma fasting triglyceride concentration (4 week value - 0 week value)
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
mg/dl | -3.5 (21.2) | 6.4 (14.0)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.11, ANCOVA; Effect of group on change of outcome with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = -7.9, 95% CI 2-sided [-17.6 to 1.8]

14. Secondary Outcome: 3-(3'-Hydroxy-4'-Methoxyphenyl)Hydracrylic
Description: Absolute change of total 24-hour urinary 3-(3'-hydroxy-4'-methoxyphenyl)hydracrylic (4 week value - 0 week value)
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
ng | 23322 (32654) | -336 (12414)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.0032, ANCOVA; Effect of group on change with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = 23340, 95% CI 2-sided [8284 to 38396]

15. Secondary Outcome: Hesperetin-3'-O-glucuronide
Description: Absolute change of total 24-hour urinary hesperetin-3'-O-glucuronide (4 week value - 0 week value)Urine concentration hesperetin-3'-O-glucuronide
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
ng | 5550 (6502) | 4 (95)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.0003, ANCOVA; Effect of group on change with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = 5558, 95% CI 2-sided [2680 to 8437]

16. Secondary Outcome: Hesperetin-3',7-0-diglucuronide
Description: Absolute change of total 24-hour urinary hesperetin-3',7-0-diglucuronide (4 week value - 0 week value)
Time Frame: 4 weeks
Population: One participant was excluded due to extreme values that deviated from the mean by more than 2 standard deviations across multiple outcomes. The exclusion was based on protocol-defined criteria. Invalid results obtained for this outcome in one participant in the sucrose group.
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 22
ng | 3797 (4955) | -3 (10)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.0012, ANCOVA; Effect of group on change with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = 3824, 95% CI 2-sided [1611 to 6036]

17. Secondary Outcome: p-Hydroxyhippuric Acid
Description: Absolute change of total 24-hour urinary p-Hydroxyhippuric acid (4 week value - 0 week value)
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
ng | 20347 (26775) | -770 (9212)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.0023, ANCOVA; Effect of group on change with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = 19522, 95% CI 2-sided [7353 to 31691]

18. Secondary Outcome: 3-(4'-Methoxyphenyl)Propionic Acid-3'-O-glucuronide
Description: Absolute change of total 24-hour urinary 3-(4'-methoxyphenyl)propionic acid-3'-O-glucuronide (4 week value - 0 week value)
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
ng | 23124 (25954) | -198 (876)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.0001, ANCOVA; Effect of group on change with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = 21881, 95% CI 2-sided [11307 to 32455]

19. Secondary Outcome: Hesperetin-7-O-glucuronide
Description: Absolute change of total 24-hour urinary hesperetin-7-O-glucuronide (4 week value - 0 week value)
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
ng | 9556 (11081) | -2 (18)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.0002, ANCOVA; Effect of group on change with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = 9666, 95% CI 2-sided [4808 to 14524]

20. Secondary Outcome: Naringin-7-O-glucuronide
Description: Absolute change of total 24-hour urinary naringen-7-O-glucuronide (4 week value - 0 week value)
Time Frame: 4 weeks
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 22
ng | 3286 (4453) | -284 (851)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.0011, ANCOVA; Effect of group on change with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = 3413, 95% CI 2-sided [1456 to 5370]

21. Secondary Outcome: Oral Glucose Tolerance Test (OGTT) Glucose 3-hour Area Under the Curve (AUC)
Description: Absolute change in OGTT 3-hour AUC glucose concentration (4-week value - 0-week value)
Time Frame: 4 week
Population: This analysis includes participants enrolled after a COVID-related protocol modification, who completed a 3-hour OGTT. These participants (n=39) did not undergo hyperinsulinemic euglycemic clamps. Final data collection and analysis for this population are complete. One participant was excluded due to extreme values that deviated from the mean by more than 2 standard deviations across multiple outcomes. The exclusion was based on protocol-defined criteria.
Measure: Mean (Standard Deviation); unit: mg/dl x 3 hours
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 21 | 17
mg/dl x 3 hours | 46.8 (56.2) | 25.6 (80.1)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.59, ANCOVA; Effect of group on change of outcome with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = 11.5, 95% CI 2-sided [-32.0 to 55.1]

22. Secondary Outcome: Oral Glucose Tolerance Test (OGTT) Insulin 3-hour Area Under the Curve
Description: Absolute change in OGTT 3-hour AUC insulin concentration (4-week value - 0-week value)
Time Frame: 4 week
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: microUnit/ml x 3 hours
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 21 | 17
microUnit/ml x 3 hours | 74.7 (114.9) | 0.1 (105.4)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.046, ANCOVA; Effect of group on change with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = 74.6, 95% CI 2-sided [1.3 to 147.9]

23. Secondary Outcome: Fasting de Novo Lipogenesis
Description: Absolute change of fasting percentage fractional rate fasting de novo lipogenesis DNL (4 week value - 0 week value)
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: %fractional rate
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
%fractional rate | 0.9 (1.8) | 0.6 (1.7)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Effect of group on change in outcome with adjustment for BMI, Outcome at baseline and gender; Test type: Superiority; p = 0.56, ANCOVA; Effect of group on change of outcome with adjustment for gender and outcome and BMI at baseline; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.7 to 1.3]

24. Other Pre Specified Outcome: Fasting Insulin
Description: Absolute change serum insulin concentration (4-week value - 0-week value)
Time Frame: 4 week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microUnit/ml
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
microUnit/ml | -0.31 (1.80) | 0.38 (2.32)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.17, ANCOVA; Effect of group on change of outcome with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = -0.80, 95% CI 2-sided [-1.94 to 0.35]

25. Other Pre Specified Outcome: Fasting Glucose
Description: Absolute change in fasting plasma glucose concentration (4-week value - 0-week value)
Time Frame: glucose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
mg/dl | 1.5 (3.8) | 0.3 (4.7)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.65, ANCOVA; Effect of group on change of outcome with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = 0.54, 95% CI 2-sided [-1.9 to 3.0]

26. Other Pre Specified Outcome: Body Weight
Description: Change in body weight (4-week value - 0-week value)
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
kg | -0.5 (1.2) | -0.5 (0.7)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.88, ANCOVA; Effect of group on change with adjustment for gender and outcome at baseline; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.5 to 0.6]

27. Other Pre Specified Outcome: Systolic Blood Pressure
Description: Change in systolic blood pressure (4-week value - 0-week value)
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
mmHg | -2.9 (10.5) | -4.2 (10.6)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.81, ANCOVA; Effect of group on change with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = 0.6, 95% CI 2-sided [-4.4 to 5.7]

28. Other Pre Specified Outcome: Diastolic Blood Pressure
Description: Change in diastolic blood pressure (4-week value minus 0-week value)
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 25 | 23
mmHg | -2.3 (7.2) | -1.0 (7.7)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.69, ANCOVA; Effect of group on change with adjustment for gender and BMI and outcome at baseline; Mean Difference (Net) = -0.7, 95% CI 2-sided [-4.4 to 2.9]

29. Other Pre Specified Outcome: Body Fat
Description: %body fat
Time Frame: 4 weeks
Population: One participant was excluded due to extreme values that deviated from the mean by more than 2 standard deviations across multiple outcomes. The exclusion was based on protocol-defined criteria. DEXA analyzer not available to scan 2 participants in orange juice group and 1 participant in sucrose group during baseline trial.
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 23 | 21
percentage of body fat | -0.9 (0.7) | -0.5 (1.0)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.10, ANCOVA; Effect of group on change of outcome with adjustment for gender and outcome at baseline; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.0 to 0.1]

30. Primary Outcome: M Value During Hyperinsulinemic Euglycemic Clamp
Description: Absolute change of M value (glucose infusion rate during final 30 minute steady state)/ fat free body mass (kg) (4 week value - 0 week value)
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: %fractional rate
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
Number analyzed (Participants) | 4 | 6
%fractional rate | -0.2 (1.9) | 0.2 (0.9)
Statistical Analysis 1: Comparison: Naturally-sweetened orange juice vs Sugar-sweetened beverage; Test type: Superiority; p = 0.55, ANCOVA; Effect of group on change of Outcome with adjustment for outcome at baseline; Mean Difference (Net) = -0.4, 95% CI 2-sided [-2.1 to 1.2]

ADVERSE EVENTS:
Time Frame: Adverse events for each participant were collected for 6 weeks.
Arm/Group | Naturally-sweetened orange juice | Sugar-sweetened beverage
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 3/25 | 0/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naturally-sweetened orange juice (N=25) | Sugar-sweetened beverage (N=24)
stomachache (Gastrointestinal disorders) | 3 (3) | 0 (0) — indigestion due to fiber or orange juice in study diet

LIMITATIONS AND CAVEATS:
It is a limitation of the trial that we did not achieve the diversity of race/ethnicity that we had planned. Due to the COVID epidemic most of our participants were University of California Davis students. Thus our demographics reflect the UC Davis student population and 63% of the participants were Asian.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT03527277/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT03527277/ICF_001.pdf